CLINICAL TRIAL: NCT01502891
Title: Translation of Comparative Effectiveness of Depression Medications Into Practice
Brief Title: Making Decisions About Depression Medications
Acronym: iADAPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Victor Montori (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Victor Montori, Professor of Medicine, Endocrinology, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 11-003507
Record Dates: First submitted 2011-12-23; First posted 2012-01-02 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Depression
Keywords: Comparative Effectiveness Research; Decision Support Techniques; Decision Making
MeSH Terms: conditions — Depression | interventions — Decision Support Techniques

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Decision aid (Active Comparator): DEPRESSION CHOICE decision aid is provided to clinician to share with patient
  Interventions: Other: Decision Aid
- Normal care (No Intervention)

INTERVENTIONS:
Other: Decision Aid — The decision aid, Depression Medication Choice, uses plain language and is designed to enhance patient understanding and satisfy the International Patient Decision Aid Standards (IPDAS) requirements for a safe and unbiased decision aid.
  Arms: Decision aid

SUMMARY:
The purpose of this study is to determine whether the Depression Medication Choice decision aid is effective in involving patients with depression in making deliberate choices when considering medication treatment.

DETAILED DESCRIPTION:
To determine the ability of decision aids to effectively translate a depression comparative effectiveness research (CER) review into practice, the investigators have developed a literacy-sensitive depression treatment decision aid, DEPRESSION MEDICATION CHOICE, which adapts the Agency for Healthcare Research and Quality (AHRQ)'s Effective Healthcare comparative effectiveness review and associated patient guide about antidepressant medicines to satisfy the needs of clinicians, patients, and other major stakeholders. The investigators will conduct a randomized study to estimate the effect of the decision aid on patient knowledge, patient involvement in decision making and decision-making quality, and on three and six-month measures of medication adherence and mental health, when compared with usual care.

ELIGIBILITY:
Inclusion Criteria:

* Presumed diagnosis of depression (PHQ-9 of 10 or greater)
* As judged by clinician, need to initiate drug treatment for depression
* Identify primary care clinician as main depression provider
* Agree to be available for follow-up survey 6 months after treatment decision

Exclusion Criteria:

* Has prior diagnosis of bipolar disorder
* Has major communication barrier (severe hearing/vision impairment, dementia, cannot communicate with clinician in same language)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2011-12; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Quality of Decision Making | Immediately following each patient's index visit and before they leave the clinic on that day, typically within 10 minutes of completing the clinical encounter.
  A modified Decisional Conflict Scale will be used to ascertain decisional quality and satisfaction with decision making. The OPTION scale will be used to assess patient involvement in decision-making by reviewing video recordings of primary care visits with inter-rater reliability. Satisfaction with decision making will be assessed also by using two specific questions that require patients to assess the extent to which they would want for themselves and recommend to others similar decision support like what they received during the visit.
Knowledge Transfer | Immediately following each patient's index visit and before they leave the clinic on that day, typically within 10 minutes of completing the clinical encounter.
  Questions have been crafted to assess knowledge about depression treatment contained in the decision aid. These questions use a response format "true/false/unsure," and are to be answered with full access to the decision aids since they are not a test of recall, but of 'use of information.'

SECONDARY OUTCOMES:
Reach and Fidelity of Use of Decision Aids | At end of study (approximately 2 years)
  Reach will be estimated by the proportion of the eligible patients who received the intervention of the entire eligible population allocated to its use. Fidelity will be determined using a checklist for each encounter to determine the proportion of visits in which more than >80% of decision aid items were delivered.
Medication Adherence to Antidepressants | Six months post-prescription
  Investigators will obtain pharmacy records to determine anti-depressant use, adherence, and persistence based on prescription refills.
Depression Control | At six months post index visit
  Investigators will assess patients at baseline, 3 and 6 months using the Patient Health Questionnaire 9 (PHQ-9) to measure the extent to which their depressed symptoms changed over time.
Clinician Satisfaction with Decision Aids | Immediately following each patient's index visit and before they leave the clinic on that day, typically within 10 minutes of completing the clinical encounter.
  Investigators will survey clinicians at the end of each index visit with a standardized clinician satisfaction questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Victor Montori, MD, Principal Investigator — Mayo Clinic
Locations (4):
- United States (4):
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Entira Family Clinics (formerly known as Family Health Services Minnesota), Saint Paul, Minnesota
  - Mayo Clinic Health System - Franciscan Healthcare, La Crosse, Wisconsin

REFERENCES:
- [Derived] Kunneman M, Branda ME, Ridgeway JL, Tiedje K, May CR, Linzer M, Inselman J, Buffington ALH, Coffey J, Boehm D, Deming J, Dick S, van Houten H, LeBlanc A, Liesinger J, Lima J, Nordeen J, Pencille L, Poplau S, Reed S, Vannelli A, Yost KJ, Ziegenfuss JY, Smith SA, Montori VM, Shah ND. Making sense of diabetes medication decisions: a mixed methods cluster randomized trial using a conversation aid intervention. Endocrine. 2022 Feb;75(2):377-391. doi: 10.1007/s12020-021-02861-4. Epub 2021 Sep 9. PMID 34499328
- [Derived] LeBlanc A, Herrin J, Williams MD, Inselman JW, Branda ME, Shah ND, Heim EM, Dick SR, Linzer M, Boehm DH, Dall-Winther KM, Matthews MR, Yost KJ, Shepel KK, Montori VM. Shared Decision Making for Antidepressants in Primary Care: A Cluster Randomized Trial. JAMA Intern Med. 2015 Nov;175(11):1761-70. doi: 10.1001/jamainternmed.2015.5214. PMID 26414670
- [Derived] LeBlanc A, Bodde AE, Branda ME, Yost KJ, Herrin J, Williams MD, Shah ND, Houten HV, Ruud KL, Pencille LJ, Montori VM. Translating comparative effectiveness of depression medications into practice by comparing the depression medication choice decision aid to usual care: study protocol for a randomized controlled trial. Trials. 2013 May 7;14:127. doi: 10.1186/1745-6215-14-127. PMID 23782672